CLINICAL TRIAL: NCT05885165
Title: Supervised Online Team-based Resistance Training Versus Unsupervised Self-administered Resistance Training for Elders: a Randomized Intervention Trial
Brief Title: Supervised Online Resistance Training vs Unsupervised Self-administered Resistance Training for Elders
Acronym: ONTRAEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Studnitz Consulting (Unknown); Aktiv Hele Livet v. Rasmus Stagsted (Unknown); Aktiv Hele Livet v. Manuel Thomasen (Unknown); Moustgaard Consulting (Unknown)
Responsible Party: Principal Investigator, Faidon Magkos, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 514-0396/23-5000
Record Dates: First submitted 2023-03-06; First posted 2023-06-01 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Healthy Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised team-based exercise (Experimental): In this arm, participants will receive guided training by an instructor in teams of 10 on the online platform Zoom.
  Interventions: Behavioral: Supervised team-based exercise
- Unsupervised exercise (Active Comparator): In this arm, participants will perform the training individually with the exercises provided on the platform Exorlive, which is a one-way communication platform. However, the first two weeks (5 training sessions) will be conducted in teams of 10 participants with the presence of an instructor who will introduce, demonstrate, and supervise correct form and technique and ensure understanding of the exercise concept.
  Interventions: Behavioral: Unsupervised exercise

INTERVENTIONS:
Behavioral: Supervised team-based exercise — The intervention is a 12-week physical exercise program with five training sessions bi-weekly lasting approximately 1 hour each.
  Arms: Supervised team-based exercise
Behavioral: Unsupervised exercise — The intervention is a 12-week physical exercise program with five training sessions bi-weekly lasting approximately 1 hour each. First two weeks are supervised, the following 10 weeks are unsupervised.
  Arms: Unsupervised exercise

SUMMARY:
The primary goal of this project is to investigate whether online supervised team-based exercise training is superior for increasing functional strength in elders compared to prescribed self-administered exercise training. Secondarily, the project aims to investigate whether adherence to online supervised team-based exercise training is greater compared to prescribed self-administered training, and if online supervised team-based exercise training can increase quality of life. Finally, this project will generate more knowledge on elderly individuals' approaches and responses to physical exercise through online services. The participants will undergo a 12-week intervention where they will be performing prescribed physical exercise for 5 hours bi-weekly and complete a 3-day dietary registration three times during the study. Participants will be randomized (2:1 ratio) to two groups and will: i) undergo supervised training in groups on an online live meeting platform by trained personnel, or ii) receive prescribed exercises through an online exercise platform but their training will be self-administered and unsupervised.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years.
* Danish reading and listening proficiency.
* Participant is in possession of either a computer, tablet, or smartphone in order to participate in Zoom meetings (supervised team-based group) or training programs via Exorlive (unsupervised group).
* The participant is able to walk independently and without external aids.

Exclusion Criteria:

* BMI > 35 kg/m2.
* Participation in other intervention studies or intention to do so, which are likely to affect the present study.
* Known diseases which may affect energy expenditure and/or satiation/satiety/food intake i.e. inflammatory bowel disease, thyroid diseases.
* Current diagnosis of eating disorder (e.g. restrained eating, disinhibition, emotional eating).
* Psychiatric disorders i.e. schizophrenia, bipolar disease or depression with hospitalization within the last 6 months.
* History or diagnosis of cardiovascular disease including current angina; myocardial infarction; coronary revascularization procedures; stroke (either ischemic or hemorrhagic, including transient ischemic attacks); symptomatic peripheral artery disease that required surgery or was diagnosed with vascular imaging techniques; ventricular arrhythmia; uncontrolled atrial fibrillation; congestive heart failure (New York Heart Association Class II to IV); myocardiopathy; and history of aortic aneurysm ≥5.5 cm in diameter or aortic aneurysm surgery within the past six months, as diagnosed by a medical doctor.
* Systolic blood pressure above 160 mmHg and/or diastolic blood pressure above 100 mmHg whether on or off treatment for hypertension. If being treated, stable treatment (i.e. no change in treatment, either dose, type of medication or other changes) within the last three months is required.
* History or diagnosis of chronic kidney disease.
* History or diagnosis of liver disease.
* Active inflammatory bowel disease, celiac disease, chronic pancreatitis or other disorder potentially causing malabsorption.
* Systemic treatment with glucocorticoids inhalations and creams etc. is allowed
* Cancer: active malignant cancer or history of malignancy within the last five years (with exception of local basal and squamous cell skin cancer).
* Previous bariatric surgery or intention to undergo bariatric surgery within the next 12 months.
* History of extensive small or large bowel resection.
* Known endocrine origin of obesity (except for treated hypothyroidism).
* Current use of prescription medication or use within the previous month that has the potential of affecting body weight such as systemic corticosteroids (excluding inhaled and topical steroids), psychoactive medication, epileptic medication, or weight loss medications (either prescription, over the counter or herbal). Low dose antidepressants are allowed if they, in the judgment of the investigator, do not affect body weight or participation in the study protocol. Levothyroxine for treatment of hypothyroidism is allowed if the subject has been on a stable dose for at least three months.
* Concurrent therapy with immunosuppressive drugs or cytotoxic agents.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in 5 times sit-to-stand | Week 0 and week 13
  Physical function, assessed by the '5 times sit-to-stand' (5xsts) test

SECONDARY OUTCOMES:
Change in 1 repetition maximum (RM) leg press | Week 0 and week 13
  Assessed on a leg press machine (Steens Physical)
Change in Fat mass | Week 0 and week 13
  Assessed by bioimpedance analysis
Change in Fat-free mass | Week 0 and week 13
  Assessed by bioimpedance analysis
Change in Resting blood pressure | Week 0 and week 13
  Measured by OMRON M2
Change in Quality of life (RAND 36-item health survey) | Week 0 and week 13
  Assessed by a 36-item short form survey questionnaire. Some questions are scored on a scale from 1-5, others from 1-2, 1-3, or 1-6. The scores are converted to values between 1-100. Some questions are reverse coded such that a high value consistently means a favorable health state.
Change in Aerobic fitness | Week 0 and week 13
  Assessed by the Åstrand-Rhymings step test
Change in Balance | Week 0 and week 13
  Assessed by the Functional Reach Test
Adherence to exercise | At every training from week 1-12
  Assessed by scoring on a Borg Rating of Perceived Exertion scale. Minimum value is 6 corresponding to resting and maximum value is 20 corresponding to maximum exertion. If any score is recorded it is interpreted as the participant having completed the training session.
Food records | Week 1, Week 6, and Week 12
  3-day dietary recall including one weekend day

CONTACTS AND LOCATIONS:
Overall Officials: Faidon Magkos, Professor, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No